CLINICAL TRIAL: NCT00579449
Title: Evaluation of a Home Visiting Program for First Time Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00014616; 5K01MH70378-3 (Other Grant/Funding Number: National Institutes of Mental Health); 6997 (Other: Duke legacy protocol number); 5K01MH070378 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Child Abuse
Keywords: child abuse; child neglect
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HF 36 (Active Comparator): For those randomly assigned to the 3-year HFD group, services begin during the third trimester of pregnancy. These families are assigned a Family Support Worker, who begins to initiate contact with the family at approximately 6 months gestation, when possible, so that the family can be engaged and services begun at seven months gestation. The Family Support Worker will provide home visiting services according the existing HFD model, which combines the empirically supported Parents as Teachers Curriculum (see attached description of the Parents as Teachers curriculum) provided in accordance with Healthy Families America standards of service delivery. The 3-year HFD group will receive services to the child's third birthday.
  Interventions: Behavioral: Healthy Families Durham
- HF 18 (Active Comparator): For those randomly assigned to the 18-month HFD group, services begin during the third trimester of pregnancy. These families are assigned a Family Support Worker, who begins to initiate contact with the family at approximately 6 months gestation, so that the family can be engaged and services begun at seven months gestation. The Family Support Worker will provide home visiting services according the existing HFD model, which combines the empirically supported Parents as Teachers Curriculum (see attached description of the Parents as Teachers curriculum) provided in accordance with Healthy Families America standards of service delivery. Services for this group are terminated when the child is 18 months old, with clinically necessary referrals made for ongoing psychosocial and health needs.
  Interventions: Behavioral: Healthy Families Durham
- YC (Active Comparator): For those assigned to the Yearly Checkup group, a clinically-trained member of the HFD team will make yearly home visits to conduct the evaluation assessment. Information about community services and assistance with referrals are provided based on needs identified.
  Interventions: Behavioral: Yearly Checkup
- MCC (No Intervention): Women placed in the community services as usual (Maternity Care Coordination only) group will receive no additional services or assessments as a part of this study.

INTERVENTIONS:
Behavioral: Healthy Families Durham — Implementation of Healthy Families America program plus Parents As Teachers curriculum
  Arms: HF 18; HF 36
Behavioral: Yearly Checkup — Mother and child are assessed annually and based on responses and stated needs, referrals to community resources are made.
  Other Names: case management
  Arms: YC

SUMMARY:
The purpose of this research is to evaluate the Healthy Families Durham (HFD) program by comparing the traditional 3-year program to 18-months of Healthy Families Durham to Yearly Visits with case management referrals to community services as usual, and to determine whether participation in the program reduces the number of reports for child maltreatment within the first seven years of the child's life.

ELIGIBILITY:
Inclusion Criteria:

* mother is a first-time parent (has been a primary caregiver of a child for less than 3 months total
* resident of Durham, North Carolina
* mother is being referred during pregnancy
* has at least one of the following risk factors: 16 years old or younger; lack of social support; history of substance abuse in the past 12 months; ever received treatment for alcohol or drug problems; history of domestic violence; history of being abused or neglected as a child; history of mental health problems in past 12 months; past child protective services involvement as a parent

Exclusion Criteria:

* actively suicidal or homicidal
* acutely psychotic
* moderately to severely mentally retarded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2005-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Durham County, North Carolina Department of Social Services reports of child maltreatment | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Robert Murphy, Ph.D., Principal Investigator — Duke University; Kenneth Dodge, Ph.D., Principal Investigator — Duke University
Locations (1):
- Center for Child and Family Health, Durham, North Carolina, United States